CLINICAL TRIAL: NCT00254826
Title: Randomized Controlled Double-Blind Trial of the Comparative Viremia, Immunogenicity and Safety of a 17-D Live Attenuated Yellow Fever Vaccine (YF-VAX)Given Alone or in Combination With Human Immune Globulin (Gama STAN S/D)
Brief Title: Yellow Fever Virus Vaccine and Immune Globulin Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mark Mulligan, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00045982
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Viremia
Keywords: Yellow Fever Virus Vaccination
MeSH Terms: conditions — Viremia | interventions — Yellow Fever Vaccine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- YF-VAX® plus saline (Other): Drug: YF-VAX® plus saline
  Interventions: Biological: YF-VAX® plus saline
- 17D YF Vaccine plus Ig (Experimental): Drug: 17D YF Vaccine plus Ig; one vaccine on day 0
  Interventions: Biological: 17D YF Vaccine plus Ig,

INTERVENTIONS:
Biological: YF-VAX® plus saline — YF-VAX® plus saine
  Arms: YF-VAX® plus saline
Biological: 17D YF Vaccine plus Ig, — 17D YF Vaccine plus Ig, one vaccine on day 0
  Arms: 17D YF Vaccine plus Ig

SUMMARY:
The purpose of this study is to determine whether immune globulin can limit the amount of yellow fever vaccine virus present in the blood after vaccination without compromising the immunity associated with the yellow fever vaccine. The study will enroll 80 participants in two groups of 40 each. The first group will receive the yellow fever vaccine with salt-water placebo. The second group will receive yellow fever vaccine with immune globulin. The amount of vaccine virus and immune response in both groups will be compared. Yellow fever vaccine has been used to protect humans against Yellow Fever Vaccine disease since the 1930s.

DETAILED DESCRIPTION:
This double-blind, randomized outpatient study is designed to determine if human immune globulin (IG) will limit the viremic response to 17D yellow fever vaccine without compromising immunogenicity. The yellow fever 17D vaccine YF-VAX® is manufactured in the United States. The IG, Gama STAN S/D®, is manufactured in the U.S. The study will be conducted in 80 healthy adults 18-40 years of age in the U.S. Participants will be randomized to receive YF-VAX® plus saline (40 subjects), or YF-VAX® plus Gama STAN S/D® (40 subjects). The dose of Gama STAN S/D® will be that used for the prevention of hepatitis A, i.e. 0.06 mL/kg. The lot of Gama STAN S/D® will have been tested and shown to contain yellow fever neutralizing antibodies at a log neutralizing index of >0.7. Saline will be given to blind the vaccine administrator and vaccinee as to their treatment group. A stratified randomization procedure will be used to ensure equal distribution of study medications to participants by gender. Safety and tolerability will be assessed by comparison of the incidence of adverse events across the two treatment groups.

The hypothesis being tested is whether co-administration of yellow fever antibody and yellow fever vaccine (passive-active immunization) results in effective immunization while reducing viremia. The effectiveness of use of Gama STAN S/D® in combination with YF-VAX® will be assessed by a reduction in the viremic response in the vaccinee. Viremia is a measure of replication of YF 17D virus in host tissues, and absence of viremia indicates that virus replication in host tissues is abrogated. Abrogation of virus replication is expected to limit the potential for dissemination of virus and virus invasion of and damage to vital organs, including the liver and brain. The methods used to quantify viremia will be reverse transcriptase-polymerase chain reaction (RT-PCR) and direct plaquing in Vero cell monolayers. In addition, sera collected pre-vaccination and on blood draws post-vaccination will be tested for yellow fever neutralizing antibodies to measure immunogenicity. The method used to detect neutralizing antibodies will be a plaque-reduction neutralization test (PRNT) performed in Vero cell culture using the constant serum-varying virus technique standardized by the U.S. Food and Drug Administration (Beaty et al., 1989). The PRNT has been recently validated and used to support Phase 3 clinical trials of YF-VAX® (Monath et al. 2002a). The primary endpoint will be the comparison of the proportion of subjects without prior yellow fever immunization in each treatment group who have measurable vaccine virus after vaccination. The T-cell activation, cytokine response, dendritic cell response and kinetics and phenotype of natural killer (NK) cells will also be characterized.

Study participants will be excluded who have significant underlying medical conditions, a history of sensitivity to IG, or established contraindications to yellow fever vaccine, including immunosuppression, thymus disorder, pregnancy, or egg hypersensitivity. These exclusion criteria represent the major contraindications to the use of Gama STAN S/D® and all yellow fever vaccines, including YF-VAX®.

The study consists of a Screening Period and a Treatment Period. During the Screening Period (Days -30 to -1), informed consent is obtained, eligibility for study entry is assessed and baseline tests are performed. Subjects who satisfy all inclusion/exclusion criteria are eligible to enter the Treatment Period and are randomized to one of the two treatment groups. On Day 0 subjects will receive either YF-VAX® plus saline, or YF-VAX® plus Gama STAN S/D®. Subjects return to the clinic for daily visits on day 1, 2, 3, 5, 7, 9, 11, 14, 30, and 91. The total duration of participation for an individual subject is approximately 91 days.

Safety assessments in vaccinated subjects include adverse event reporting and clinical laboratory evaluations. To ensure thorough reporting of adverse events during the time interval in which adverse events associated with yellow fever vaccination might be expected to occur, subjects will be required to complete a study diary for Days 0-28. The study diary will record both local reactions (i.e., pain, redness, and swelling) and systemic reactions (i.e., feeling ill [malaise], headache, muscle aches, fever, chills, rash, tiredness, and other general symptoms). These are the principal symptoms and side effects known to be associated with yellow fever 17D vaccine. At each visit, study personnel will perform clinical evaluations and at days 7, 14 and 30 the study staff will review the diary card and follow up on any adverse events that occurred since vaccination.

A sample size for efficacy of 80 participants including 40 subjects in the group receiving YF-VAX® plus saline and 40 subjects receiving YF-VAX® plus Gama STAN S/D® provides 80% power in a one-sided test at significance level alpha of 0.05, assuming 93% of subjects not receiving immune globulin will exhibit detectable viremia and a reduction of 35% (to 61% of subjects) following administration of immune globulin.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and give informed consent
* Age 18-40 years old
* No medical contraindications to participation discovered at the screening visit
* Negative serologic test for HIV, HCV and Hepatitis B surface antigen at the screening visit
* Female volunteers of childbearing potential must agree to use effective birth control throughout the duration of the study. A negative urine pregnancy test must be documented prior to any injection.
* Must weigh at least 110 lbs

Exclusion Criteria:

* Any history of allergy or history of anaphylaxis to any of the vaccine components
* Any history of allergic reaction to human immune globulin or a history of IgA deficiency
* History of hypersensitivity to ingestion of eggs or allergic reaction to vaccines prepared in eggs or chick embryo cell cultures (e.g. influenza, measles)
* Known or suspected immunodeficiency (e.g. HIV infection, primary immunodeficiency disorder, leukemia, lymphoma), use of immunosuppressive or antineoplastic drugs (corticosteroids> 10 mg prednisolone/prednisone, or equivalent, for mare than 14 days in the last three months). Persons with previous skin cancer or cured non-lymphatic tumors are not excluded from the study.
* Any clinically significant chronic medical condition that is considered progressive including: hypertension, diabetes, gastrointestinal abnormalities (e.g. active peptic ulcer disease), cardiac, pulmonary, hepatic, renal, or neurologic disease.
* History of excessive alcohol consumption, drug abuse, psychiatric conditions, social conditions, or occupational requirements that in the opinion of the investigator would preclude compliance with the trial
* Receipt of any live or inactivated vaccine between the screening visit and the day 0 visit, or any vaccine within 30 days of a vaccination visit
* Any subject found to be HIV positive, hepatitis B surface antigen positive, or hepatitis C antibody positive at the time of screening
* Any contraindication to intramuscular injection
* Women who are pregnant, nursing or expect to become pregnant during the study period
* Administration of a blood product or immune globulin product within 6 months of injection
* History of previous yellow fever, West Nile, dengue, St. Louis encephalitis, Japanese encephalitis or tick-borne encephalitis vaccination or infection
* Serologic evidence of previous yellow fever, West Nile, dengue, St. Louis encephalitis, Japanese encephalitis or tick-borne encephalitis vaccination or infection
* History of travel to a yellow fever endemic zone as defined by the Centers for Disease Control and Prevention. Health Information for International Travel, 2005-2006
* History of thymus disorder or dysfunction, including myasthenia gravis, thymoma, thymectomy, or DiGeorge syndrome
* History of an autoimmune disorder

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2006-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Compare the proportion of participants developing viremia between the group receiving the yellow fever vaccine/saline and yellow fever vaccine with human immune globulin. | 91 Days

SECONDARY OUTCOMES:
Compare the viremia levels between the group of vaccinees receiving yellow fever vaccine with the group receiving yellow fever vaccine with human immune globulin. | 91 days
Compare the dynamics of T cell activation, cytokine response and dendritic cell response in vaccinees during primary response to yellow fever vaccine to vaccinees given yellow fever vaccine given in combination with human immune globulin. | 91 days
Compare the geometric mean neutralizing antibody titer in the group of yellow fever vaccinees with the group of vaccinees receiving yellow fever vaccine in combination with human immune globulin. | 91 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark J. Mulligan, MD, Principal Investigator — Emory University
Locations (1):
- Emory Vaccine Center-The Hope Clinic and The Pediatric ID Clinic, Decatur, Georgia, United States

REFERENCES:
- [Derived] Edupuganti S, Eidex RB, Keyserling H, Akondy RS, Lanciotti R, Orenstein W, del Rio C, Pan Y, Querec T, Lipman H, Barrett A, Ahmed R, Teuwen D, Cetron M, Mulligan MJ; YF-Ig Study Team. A randomized, double-blind, controlled trial of the 17D yellow fever virus vaccine given in combination with immune globulin or placebo: comparative viremia and immunogenicity. Am J Trop Med Hyg. 2013 Jan;88(1):172-7. doi: 10.4269/ajtmh.2012.12-0179. Epub 2012 Dec 3. PMID 23208880
- See also: Emory Vaccine Center-The Hope Clinic — http://www.hopeclinic.emory.edu